CLINICAL TRIAL: NCT04474548
Title: Postplacental LNG-IUD Ultrasound Use Study
Acronym: PLUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20D.502
Record Dates: First submitted 2020-07-13; First posted 2020-07-17 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: IUD Insertion Complication
Keywords: IUD; Postpartum; Ultrasound

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound (Experimental): For participants randomly assigned to ultrasound use, a bedside ultrasound will be performed using the trans-abdominal probe during and/or immediately after placement of the IUD. The distance from the IUD arms to the fundus will be measured with the ultrasound, and the IUD will be defined as being "in place" when the distance from the top of the IUD to the fundus is measured to be 3mm or less. If the distance is greater than 4mm, the provider may reposition the IUD manually or with a ring forceps.
  Interventions: Other: Ultrasound use
- No ultrasound (No Intervention): For participants randomly assigned to no ultrasound use, provider will insert the IUD with a ring forceps and will use palpation of the fundus to determine whether or not the IUD is likely in place.

INTERVENTIONS:
Other: Ultrasound use — Ultrasound will be used to determine location of IUD after insertion.
  Arms: Ultrasound

SUMMARY:
This study will enroll women planning to have an intrauterine device (IUD) placed for contraception immediately following a vaginal delivery. Women will be randomized to have this procedure done with or without ultrasound guidance. We intend to determine if the routine use of ultrasound to confirm device position reduces the rates of IUD expulsion.

DETAILED DESCRIPTION:
Participants will be screened and consented for participation in the study when they are admitted to Labor and Delivery for delivery and express desire for a post-placental LNG-IUD. If the patient consents for study participation and meets eligibility criteria above, she will be enrolled in the study after achieving vaginal delivery when she is randomized to either IUD insertion with ultrasound or without ultrasound use. See protocol for detailed description of IUD placement and ultrasound use.

After placement of IUD with or without ultrasound guidance, patients will be scheduled for a routine postpartum follow-up visit 6-10 weeks after delivery. At the postpartum follow-up visit, providers will assess for IUD expulsion with usual clinical practice, including history, pelvic exam, and additional imaging if IUD strings are not visualized on exam. Several attempts to contact participants who do not attend their postpartum visits will be made to attempt to reschedule appointments and conduct a phone questionnaire assessing for IUD expulsion.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to Thomas Jefferson University Labor and Delivery who desire and consent to post-placental LNG-IUD placement
* English- and Spanish- speaking patients

Exclusion Criteria:

* Patients undergoing planned or unplanned Cesarean delivery
* Patients who have an allergy or other contraindication to use of LNG-IUD
* Patients who tested positive for gonorrhea or chlamydia during pregnancy without treatment and a subsequent negative test of cure
* Patients with one or more leiomyomata greater than 3 cm in diameter impinging the uterine cavity
* Clinical diagnosis of chorioamnionitis or presumed chorioamnionitis in labor
* Postpartum hemorrhage as defined by need for transfusion, estimated blood loss greater than 1000mL, or use of 3 or more doses of uterotonic medications

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
IUD expulsion | 6-10 weeks
  The primary objective is to determine whether the expulsion rate of the LNG-releasing IUD within a 6-10 week period would be different when inserted with ultrasound guidance or with no ultrasound confirmation

SECONDARY OUTCOMES:
IUD insertion complication | 6-10 weeks
  To determine if rate of complication with insertion, such as uterine perforation rates, infection rates, or bleeding rates, are different with or without ultrasound guidance
Receiving IUD | 6-10 weeks
  To determine what percentage of patients who desire a post-placental IUD after delivery are able to receive one and to determine if enrolled patients that cannot get an immediate post-placental IUD get an IUD within 6-10 weeks after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Perriera, MD, MPH, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No